CLINICAL TRIAL: NCT03742895
Title: A Phase 2 Study of Olaparib Monotherapy in Participants With Previously Treated, Homologous Recombination Repair Mutation (HRRm) or Homologous Recombination Deficiency (HRD) Positive Advanced Cancer
Brief Title: Efficacy and Safety of Olaparib (MK-7339) in Participants With Previously Treated, Homologous Recombination Repair Mutation (HRRm) or Homologous Recombination Deficiency (HRD) Positive Advanced Cancer (MK-7339-002 / LYNK-002)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7339-002; MK-7339-002 (Other: MSD Protocol Number); LYNK-002 (Other: MSD); 194694 (Registry Identifier: JAPIC-CTI); 2018-003007-19 (EudraCT Number)
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Neoplasms
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Participants with HRRm or HRD-positive advanced cancer will receive oral olaparib, 300 mg twice daily (BID).
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib 300 mg administered BID as two, 150 mg oral tablets.
  Other Names: MK-7339; AZD2281; KU-0059436; LYNPARZA®

SUMMARY:
This study will evaluate the efficacy and safety of olaparib (MK-7339) monotherapy in participants with multiple types of advanced cancer (unresectable and/or metastatic) that: 1) have progressed or been intolerant to standard of care therapy; and 2) are positive for homologous recombination repair mutation (HRRm) or homologous recombination deficiency (HRD).

ELIGIBILITY:
Inclusion Criteria:

* For all participants:
* Has measurable disease per RECIST 1.1 or PCWG-modified RECIST 1.1 as assessed by the local site Investigator/radiology and confirmed by BICR.
* Is able to provide a newly obtained core or excisional biopsy of a tumor lesion or either an archival formalin-fixed paraffin embedded (FFPE) tumor tissue block or slides.
* Has a life expectancy of at least 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1, as assessed within 7 days of treatment initiation.
* Male participants must agree to use contraception during the treatment period and for at least 95 days (3 months and 5 days) after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  1. Is not a woman of childbearing potential (WOCBP).
  2. Is a WOCBP and using a contraceptive method that is highly effective with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 180 days after the last dose of study intervention, AND agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period. Abstains from breastfeeding during the study intervention period and for at least 30 days after the last dose of study intervention.
* Has adequate organ function.
* For participants who have non-breast or -ovarian cancers that are breast cancer susceptibility gene 1/2 (BRCA1/2) mutated (BRCAm), or who have cancers that are BRCA1/2 non-mutated and homologous recombination repair nonmutated:
* Has a histologically- or cytologically-confirmed advanced (metastatic and/or unresectable) solid tumor (except ovarian cancer whose tumor has a germline or somatic BRCA mutation and breast cancer whose tumor has a germline BRCA mutation) that is not eligible for curative treatment and for which standard of care therapy has failed. Participants must have progressed on or be intolerant to standard of care therapies that are known to provide clinical benefit. There is no limit on the number of prior treatment regimens.
* Has either centrally-confirmed known or suspected deleterious mutations in at least 1 of the genes involved in HRR or centrally-confirmed HRD.
* For participants receiving prior platinum (cisplatin, carboplatin, or oxaliplatin either as monotherapy or in combination) for advanced (metastatic and/or unresectable) solid tumor, have no evidence of disease progression during the platinum chemotherapy or ≤4 weeks of completing the platinum-containing regimen.
* For participants who have somatic BRCAm breast cancer:
* Has histologically- or cytologically-confirmed breast cancer with evidence of metastatic disease.
* Has a known or suspected deleterious mutation in breast cancer susceptibility gene (BRCA) 1 or BRCA2 and does not harbor a germline BRCA1 or BRCA2 mutation - testing can be done centrally or locally. Blood and tissue samples must be provided by all participants.
* Has received treatment with an anthracycline unless contraindicated and a taxane in either the neoadjuvant/adjuvant or metastatic setting.
* Participants with estrogen and/or progesterone receptor-positive disease must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy.

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, ductal carcinoma in situ, or cervical carcinoma in situ that has undergone potentially curative therapy are not excluded.
* Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Participants with previously treated brain metastases may participate if radiologically stable, clinically stable, and without requirement for steroid treatment for at least 14 days prior to the first dose of study treatment.
* Has received colony-stimulating factors (e.g., granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study treatment.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active hepatitis infection (i.e., Hepatitis B or C).
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (e.g., gastrectomy, partial bowel obstruction, malabsorption).
* Has received prior therapy with olaparib or with any other polyadenosine 5' diphosphoribose (poly[ADP ribose]) polymerization (PARP) inhibitor.
* Has a known hypersensitivity to the components or excipients in olaparib.
* Has received previous allogenic bone-marrow transplant or double umbilical cord transplantation (dUCBT).
* Has received a whole blood transfusion in the last 120 days prior to entry to the study. Packed red blood cells and platelet transfusions are acceptable if not performed within 28 days of the first dose of study treatment.
* Has received any anti-neoplastic systemic chemotherapy or biological therapy, targeted therapy, or an anticancer hormonal therapy within 3 weeks prior to the first dose of study intervention.
* Has a primary cancer of unknown origin.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 53 months
  ORR is defined as the percentage of participants who achieve a confirmed complete response ([CR]; disappearance of all target lesions) or partial response ([PR]: ≥30% decrease in the sum of diameters of target lesions) as assessed by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors 1.1, modified to follow a maximum of 10 target lesions in total and a maximum of 5 target lesions per organ (modified RECIST 1.1). For participants with prostate cancer, ORR will be based on Prostate Cancer Working Group (PCWG)-modified RECIST 1.1 as assessed by BICR.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 53 months
  DOR is defined as the time from first documented evidence of CR or PR until the first documented sign of disease progression or death due to any cause, whichever occurs first. DOR will be assessed by BICR according to either modified RECIST 1.1 or PCWG-modified RECIST 1.1 for participants with prostate cancer.
Overall Survival (OS) | Up to 53 months
  OS is defined as the time from the date of the first dose to the date of death due to any cause.
Progression Free Survival (PFS) | Up to 53 months
  PFS is defined as the time from the date of the first dose to either: 1) the first documented disease progression as assessed either by BICR according to modified RECIST 1.1 or PCWG-modified RECIST 1.1 for participants with prostate cancer; or 2) death due to any cause, whichever occurs first.
Number of Participants Experiencing an Adverse Event (AE) | Up to 53 months
  An AE is any unfavorable and unintended sign, symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing an AE will be assessed.
Number of Participants Discontinuing Study Treatment due to an Adverse Event (AE) | Up to 52 months
  The number of participants discontinuing study treatment due to an AE will be assessed.
Objective Response Rate (ORR) in Participants with HRRm or HRD Positive Cancer | Up to 53 months
  For participants with homologous recombination repair mutation (HRRm) or homologous recombination deficiency (HRD) positive cancer, the ORR will be assessed. ORR is defined as the percentage of participants who achieve a confirmed complete response ([CR]; disappearance of all target lesions) or partial response ([PR]: ≥30% decrease in the sum of diameters of target lesions) as assessed by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors 1.1, modified to follow a maximum of 10 target lesions in total and a maximum of 5 target lesions per organ (modified RECIST 1.1). For participants with prostate cancer, ORR will be based on Prostate Cancer Working Group (PCWG)-modified RECIST 1.1 as assessed by BICR.
Time to Earliest Progression by Cancer Antigen-125 (CA-125) | Up to 53 months
  For participants with BRCA1/2 non-mutated ovarian cancer only, the time to earliest progression by CA-125 will be assessed. Progression by CA-125 is defined as an increase in CA-125 level ≥2x upper limit normal (ULN) on 2 occasions, 1 week apart. For participants with elevated CA-125 (≥ULN) at baseline, progression by CA-125 is defined as an increase in CA-125 level ≥2x the nadir value on 2 occasions, 1 week apart.
Prostate-specific Antigen (PSA) Response Rate in Participants with Prostate Cancer | Up to 53 months
  For participants with prostate cancer, the PSA response rate will be presented. PSA response rate is defined as the percentage of participants in the analysis population with PSA reduction of ≥50% from baseline measured twice at least 3 weeks apart.
Progression-Free Survival After Next-Line Treatment in Participants with sBRCAm Breast Cancer | Up to 53 months
  For participants with somatic BRCA mutated (sBRCAm) breast cancer, the PFS after next-line treatment will be presented. PFS is defined as the time from the date of the first dose to either: 1) the first documented disease progression on the next-line of treatment, as assessed by BICR according to modified RECIST 1.1; or 2) death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (130):
- United States (24):
  - The University of Arizona Cancer Center - North Campus ( Site 0011), Tucson, Arizona
  - St Joseph Heritage Healthcare-Oncology ( Site 0056), Fullerton, California
  - Cedars Sinai Medical Center ( Site 0002), Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center ( Site 0007), San Francisco, California
  - Rocky Mountain Regional Veterans Affairs Medical Center ( Site 0092), Aurora, Colorado
  - Winship Cancer Institute of Emory University ( Site 0025), Atlanta, Georgia
  - Augusta University ( Site 0028), Augusta, Georgia
  - Markey Cancer Center ( Site 0018), Lexington, Kentucky
  - University of Maryland ( Site 0050), Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square ( Site 0054), Baltimore, Maryland
  - University of Massachusetts ( Site 0017), Worcester, Massachusetts
  - Henry Ford Health System ( Site 0060), Detroit, Michigan
  - Cancer Partners of Nebraska ( Site 0051), Lincoln, Nebraska
  - Memorial Sloan Kettering Cancer Center- Monmouth ( Site 0116), Middletown, New Jersey
  - Memorial Sloan-Kettering Cancer Center at West Harrison ( Site 0126), Harrison, New York
  - VA New York Harbor Healthcare System Manhattan ( Site 0094), New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0057), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0026), New York, New York
  - Southwestern Regional Medical Center, Inc. ( Site 0079), Tulsa, Oklahoma
  - Eastern Regional Medical Center, Inc. ( Site 0077), Philadelphia, Pennsylvania
  - Sanford Hematology Oncology-Sioux Falls SD ( Site 0012), Sioux Falls, South Dakota
  - Intermountain Healthcare ( Site 0043), St. George, Utah
  - Virginia Mason Medical Center ( Site 0052), Seattle, Washington
  - Veterans Affairs Puget Sound Health Care System [Seattle, WA] ( Site 0093), Seattle, Washington
- Argentina (4):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 2703), Berazategui, Buenos Aires
  - Hospital Britanico de Buenos Aires ( Site 2704), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Instituto de Investigaciones Metabolicas ( Site 2700), Buenos Aires
  - Hospital Aleman ( Site 2702), Buenos Aires
- Australia (3):
  - Kinghorn Cancer Centre ( Site 2200), Darlinghurst, New South Wales
  - MNCCI Port Macquarie Base Hospital ( Site 2201), Port Macquarie, New South Wales
  - Linear Clinical Research Ltd ( Site 2202), Nedlands, Western Australia
- Canada (4):
  - Sunnybrook Research Institute ( Site 0210), Toronto, Ontario
  - Hopital Maisonneuve-Rosemont CIUSSS de l Est de L Ile de Montreal ( Site 0203), Montreal, Quebec
  - Jewish General Hospital ( Site 0209), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- Colombia (9):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 2812), Medellín, Antioquia
  - Rodrigo Botero SAS ( Site 2801), Medellín, Antioquia
  - Biomelab S A S ( Site 2800), Barranquilla, Atlántico
  - Administradora Country SA - Clinica del Country ( Site 2802), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 2807), Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerologia E.S.E ( Site 2809), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 2808), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 2806), Montería, Departamento de Córdoba
  - C. Medico Imbanaco Cali S.A. ( Site 2810), Cali, Valle del Cauca Department
- Denmark (3):
  - Rigshospitalet ( Site 0402), Copenhagen, Capital Region
  - Herlev og Gentofte Hospital. ( Site 0401), Herlev, Capital Region
  - Odense Universitetshospital ( Site 0400), Odense, Region Syddanmark
- France (6):
  - CHU Poitiers ( Site 0612), Poitiers, Ain
  - Centre Antoine Lacassagne ( Site 0610), Nice, Alpes-Maritimes
  - Institut de Cancerologie Strasbourg Europe ( Site 0613), Strasbourg, Alsace
  - Centre Georges Francois Leclerc ( Site 0608), Dijon, Bourgogne-Franche-Comté
  - Institut Bergonie ( Site 0603), Bordeaux, Gironde
  - Institut Gustave Roussy ( Site 0601), Villejuif, Val-de-Marne
- Guatemala (4):
  - Centro Regional de Sub Especialidades Medicas SA ( Site 3003), Guatemala, Departamento de Quetzaltenango
  - Centro de Investigaciones Clinicas de Latinoamerica S.A. - CELAN ( Site 3004), Guatemala City
  - Integra Cancer Institute ( Site 3006), Guatemala City
  - Grupo Angeles SA ( Site 3001), Guatemala City
- Ireland (4):
  - Mater Misericordiae University Hospital ( Site 1654), Dublin, Carlow
  - Bon Secours Hospital ( Site 1656), Cork
  - St. Vincent's University Hospital ( Site 1653), Dublin
  - Tallaght University Hospital ( Site 1652), Dublin
- Israel (5):
  - Soroka Medical Center ( Site 0800), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0801), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0802), Jerusalem
  - Chaim Sheba Medical Center ( Site 0803), Ramat Gan
  - Sourasky Medical Center ( Site 0804), Tel Aviv
- Italy (3):
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 0700), Napoli, Campania
  - Istituto Clinico Humanitas Research Hospital ( Site 0703), Rozzano, Lombardy
  - Policlinico Le Scotte di Siena ( Site 0704), Siena, Tuscany
- Japan (6):
  - Aichi Cancer Center Hospital ( Site 2602), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2600), Kashiwa, Chiba
  - Kyoto University Hospital ( Site 2603), Kyoto, Kyoto
  - Osaka University Hospital ( Site 2604), Suita, Osaka
  - National Cancer Center Hospital ( Site 2601), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2605), Tokyo
- Mexico (8):
  - Actualidad Basada en la Investigacion del Cancer ( Site 2903), Guadalajara, Jalisco
  - Unidad Biomedica Avanzada Monterrey S. A. ( Site 2902), Monterrey, Nuevo León
  - Cuidados Oncologicos ( Site 2908), Santiago de Quetaro, Querétaro
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares ( Site 2901), Madero, Tamaulipas
  - Centro Estatal de Cancerologia de Chihuahua ( Site 2907), Chihuahua City
  - CRYPTEX Investigacion Clinica S.A. de C.V. ( Site 2900), Mexico City
  - CENEIT Oncologicos ( Site 2904), México
  - Oaxaca Site Management Organization S.C. ( Site 2905), Oaxaca City
- Peru (9):
  - Hospital de Alta Complejidad de La Libertad Virgen de La Puerta ( Site 3102), Trujillo, La Libertad
  - Instituto Nacional de Enfermedades Neoplasicas ( Site 3106), Lima, Muni Metro de Lima
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 3107), Lima
  - Clinica Internacional Sede San Borja ( Site 3100), Lima
  - Instituto de Oncologia y Radioterapia Clinica Ricardo Palma ( Site 3101), Lima
  - Oncosalud-Clinical Research ( Site 3108), Lima
  - Hospital Central de la Fuerza Aerea del Peru ( Site 3104), Lima
  - Hospital Militar Central Coronel Luis Arias Schereiber ( Site 3105), Lima
  - Hospital Arzobispo Loayza ( Site 3103), Lima
- Romania (7):
  - S.C. Pelican Impex S.R.L Spitalul Clinic Pelican Oradea ( Site 1102), Oradea, Bihor County
  - Medisprof ( Site 1107), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL ( Site 1105), Comuna Floresti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 1103), Craiova, Dolj
  - Spitalul PDR Medlife ( Site 1106), Brasov
  - S.C.Focus Lab Plus S.R.L ( Site 1101), Bucharest
  - S.C.Gral Medical S.R.L ( Site 1104), Bucharest
- Russia (11):
  - Arkhangelsk Clinical Oncological Dispensary ( Site 1204), Arkhangelsk, Arkhangelskaya oblast
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 1212), Chelyabinsk, Chelyabinsk Oblast
  - N.N. Blokhin NMRCO ( Site 1201), Moscow, Moscow
  - MSROI named after P.A. Hertsen branch of FSBI NMRC Radiology ( Site 1213), Moscow, Moscow
  - MEDSI Clinical Hospital on Pyatnitsky Highway-Departmentof Antitumor Drug therapy ( Site 1216), Krasnogorsk, Moscow Oblast
  - Ryazan Regional Clinical Oncology dispensary ( Site 1202), Ryazan, Ryazan Oblast
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 1211), Samara, Samara Oblast
  - Clinical Hospital Saint Luka ( Site 1205), Saint Petersburg, Sankt-Peterburg
  - SBHI Leningrad Regional Clinical Hospital ( Site 1206), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1208), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH named after professor M.Z. Sigal ( Site 120, Kazan', Tatarstan, Respublika
- South Korea (3):
  - Seoul National University Bundang Hospital ( Site 2402), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 2401), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2400), Seoul
- Spain (2):
  - Hospital Universitario Quiron Madrid ( Site 1352), Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d Hebron ( Site 1350), Barcelona
- Switzerland (3):
  - Universitaetsspital Zuerich ( Site 1400), Zuerich, Canton of Aargau
  - Hopitaux Universitaires de Geneve HUG. ( Site 1406), Geneva, Canton of Geneva
  - Ospedale Regionale di Bellinzona e Valli ( Site 1407), Bellinzona, Canton Ticino
- Turkey (Türkiye) (8):
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi ( Site 1507), Konya, Adana
  - Baskent University Adana Training Hospital ( Site 1508), Adana
  - Hacettepe Universitesi Tıp Fakultesi ( Site 1503), Ankara
  - Akdeniz Universitesi Tip Fakultesi ( Site 1504), Antalya
  - Trakya Universitesi Tip Fakultesi ( Site 1500), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 1505), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 1506), Istanbul
  - Ege Universitesi Tip Fakultesi ( Site 1502), Izmir
- United Kingdom (4):
  - Churchill Hospital ( Site 1606), Oxford, Worcestershire
  - Christie NHS Foundation Trust ( Site 1601), Manchester
  - Northern Centre for Cancer Care ( Site 1602), Newcastle upon Tyne
  - Weston Park Hospital ( Site 1607), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26194&tenant=MT_MSD_9011